CLINICAL TRIAL: NCT04051294
Title: A Clinical Trial to Measure the Biochemical Response of Kombucha Tea in Humans
Brief Title: The Effect of Kombucha on Blood Sugar Levels in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Julie Kapp, Associate Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2014707
Record Dates: First submitted 2019-08-07; First posted 2019-08-09 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Glucose; Glucose Metabolism Disorders (Including Diabetes Mellitus); Blood Sugar; High
Keywords: kombucha; kombucha tea; tea; fermented food
MeSH Terms: conditions — Glucose Metabolism Disorders; Hyperglycemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention group 1: commercial kombucha (Experimental): 8oz
  Interventions: Dietary Supplement: Commercial kombucha tea
- Intervention group 2: brewed kombucha (Experimental): 8oz
  Interventions: Dietary Supplement: Brewed kombucha tea
- Control group 1: tea (Active Comparator): 8oz
  Interventions: Other: Control: Tea
- Control group 2: water (Placebo Comparator): 8oz
  Interventions: Other: Control: Water

INTERVENTIONS:
Dietary Supplement: Commercial kombucha tea — Commercially-available kombucha tea.
  Arms: Intervention group 1: commercial kombucha
Dietary Supplement: Brewed kombucha tea — Kombucha tea brewed
  Arms: Intervention group 2: brewed kombucha
Other: Control: Tea — Tea brewed in our lab.
  Arms: Control group 1: tea
Other: Control: Water — Tap water
  Arms: Control group 2: water

SUMMARY:
As a phase 0 clinical trial, we will learn how kombucha influences glucose metabolism in humans.

DETAILED DESCRIPTION:
Consumption of kombucha, a fermented tea beverage, has been promoted for a wide range of health benefits. However, a systematic literature review (Kapp & Sumner, 2019) revealed a lack of evidence for human health benefit. Despite the lack of evidence, U.S. retail sales of kombucha and other fermented beverages have increased 37.4% in 2017, and kombucha is the fastest growing product in the functional beverage market.

As a phase 0 clinical trial, we will learn how kombucha influences glucose metabolism in humans. We plan for 20 subjects to take part in this study.

This is a randomized-controlled counter-balanced study design. Subjects will be asked to complete 4 in-person visits over 2 months time (twice per month). At the first visit, subjects will be randomized into one of four groups. At each subsequent visit, subjects will be randomized into one of the remaining groups until they have completed each arm.

Arms (at least 5 subjects in each arm, minimum total=20 subjects)

1. Intervention group 1: commercial kombucha: drink 8oz kombucha
2. Intervention group 2: brewed kombucha: drink 8oz kombucha
3. Control group: drink 8oz tea (the same type as used to brew the kombucha)
4. Control group 2: drink 8oz tap water

ELIGIBILITY:
Inclusion Criteria:

* Men or women ages 30-65 years old
* English-speaking
* Have transportation to campus
* Overweight (BMI >= 25 kg/m2) or obese (BMI >=30 kg/m2)

Exclusion Criteria:

* Currently use any type of nicotine product
* A diagnosis of any of the following:

  * Diabetes (type 1 or 2)
  * Cancer
  * COPD
  * Chronic alcoholism
  * Peripheral vascular disease
  * Autoimmune disease
  * Chronic kidney disease
* Pregnant or breastfeeding
* Prescribed medication for insulin, glucose-lowering drugs, or steroids, such as prednisone
* Have routinely taken prebiotic or probiotic supplements in the past 3 months
* Have routinely consumed any of the following more than one time per week in the past month: kombucha, kefir, yogurt, kimchi, cottage cheese, raw apple cider vinegar (with the "mother"), sauerkraut, kvass.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Fasting blood glucose level | Baseline
  Blood drawn following a 10-12 hour fast.
Fasting insulin level. | Baseline
  Blood drawn following a 10-12 hour fast.
Blood glucose level | 3 hour
  Oral glucose tolerance test
Insulin level | 3 hour
  Oral glucose tolerance test

SECONDARY OUTCOMES:
Blood pressure | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Kapp, MPH, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States